CLINICAL TRIAL: NCT01829880
Title: Impact of Body Composition Changes and Cachexia on Bisoprolol and Ramipril Pharmacokinetics and Renal Function Estimation in Patients With Chronic Heart Failure
Brief Title: Impact of Body Composition on Bisoprolol and Ramipril Pharmacokinetics in Patients With Chronic Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University Clinic of Pulmonary and Allergic Diseases Golnik (Other)
Responsible Party: Principal Investigator, Mitja Lainščak, MD, PhD, The University Clinic of Pulmonary and Allergic Diseases Golnik
Other Study IDs: GOLNIK_PKT1
Record Dates: First submitted 2013-04-08; First posted 2013-04-11 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Chronic Heart Failure; Cachexia
Keywords: Chronic heart failure; Bisoprolol; Ramipril; Pharmacokinetic; Cachexia; Body composition; Renal function; Iohexol
MeSH Terms: conditions — Cachexia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, serum

GROUPS / COHORTS (1):
- Chronic heart failure patients: Patients with chronic heart failure who attend to internal medicine outpatient clinic.

SUMMARY:
The purpose of this study is to determine if cachexia and changes in body composition influence pharmacokinetics of bisoprolol and ramipril and the accuracy of equations for renal function estimation.

DETAILED DESCRIPTION:
Patients with chronic heart failure on treatment with bisoprolol and/or ramipril will be included. Study will consist of two study visits: baseline visit (V1) and visit which will be performed at least 6 months after baseline (V2). At both visits same procedures will be performed. On the day of the visit, patients will be asked to take their morning dose of bisoprolol and/or ramipril after the withdrawal of the first morning plasma sample. Additional 3 to 5 plasma samples will be taken within 5 hours post bisoprolol and/or ramipril dose in order to determine pharmacokinetic profile of both drugs. Body composition will be measured by bioimpedance and dual-energy X-ray absorptiometry. Renal function will be measured by clearance of intravenously administered iohexol. Biochemical parameters, muscle strength, fatigue and anorexia will be assessed in order to determine presence of cachexia.

Changes in body composition will be correlated with changes in pharmacokinetic parameters of bisoprolol and ramipril. Pharmacokinetic parameters in cachectic patients will be compared to pharmacokinetic parameters in non-cachectic patients. Parameters of body composition will be correlated with the difference between measured and estimated renal function.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic heart failure of New York Heart Association Functional Classification (NYHA) class II and III
* On treatment with bisoprolol for at least 3 days and/or ramipril for at least 4 days before V1
* Able and willing to provide freely given written informed consent

Exclusion Criteria:

* Chronic renal disease with estimated glomerular filtration rate calculated by Modification of Diet in Renal Disease (MDRD) equation < 40 mL/(min x 1,73 m2) at V1 or V2
* Liver disease or increased serum liver enzymes (bilirubin > 1.5 x normal, gamma-glutamyl transpeptidase (GGT) > 2.5 x normal, aspartate transaminase (AST) > 2.5 x normal, alanine transaminase (ALT) > 2.5 x normal) at V1 or V2
* Absence of bisoprolol or ramipril steady state concentrations at V1 or V2 or withdrawal of bisoprolol and/or ramipril in-between both visits
* Acute decompensation of heart failure in less than 4 weeks before V1 or V2
* Addition, withdrawal or change in dose of drugs that importantly influence bisoprolol or ramipril pharmacokinetics in-between V1 and V2
* Unable to understand and comply with protocol or to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic heart failure who attend internal medicine outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-07 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of bisoprolol and ramipril | Baseline and 6 months
  Pharmacokinetic parameters of bisoprolol and ramipril(clearance, volume of distribution, area under concentration-time curve, maximal concentration, time to maximal concentration) will be determined. The relation between pharmacokinetic parameters and body composition/cachexia will be assessed.

SECONDARY OUTCOMES:
Body composition | Baseline and 6 months
  Body composition (percentage and amount of body fat, lean body mass, dry lean body mass and body water) will be measured by bioimpedance and dual energy X-ray absorptiometry
Cachexia diagnosis | Baseline and 6 months
  Cachexia diagnosis (determination of low body mass index, wasting, biochemical parameters, muscle strength, fatigue and anorexia)
Renal function | Baseline and 6 months
  Renal function will be measured by clearance of intravenously applied iohexol. Estimation of renal function will be calculated with different equations based on serum creatinine concentration. Measured and estimated renal function will be compared and the differences related to body composition parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Mitja Lainscak, MD, PhD, Study Chair — University Clinic Golnik
Locations (1):
- University Clinic of Respiratory and Allergic Diseases Golnik, Golnik, Slovenia

REFERENCES:
- [Derived] Cvan Trobec K, Kerec Kos M, von Haehling S, Anker SD, Macdougall IC, Ponikowski P, Lainscak M. Iohexol clearance is superior to creatinine-based renal function estimating equations in detecting short-term renal function decline in chronic heart failure. Croat Med J. 2015 Dec;56(6):531-41. doi: 10.3325/cmj.2015.56.531. PMID 26718759